CLINICAL TRIAL: NCT04012359
Title: Lung Ultrasound Characterization of Bullous Emphysema
Brief Title: Description of Bullous Emphysema Using Lung Ultrasound and Comparison to the Characteristics of Pneumothorax
Acronym: BulleEcho
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/006/OB
Record Dates: First submitted 2019-05-24; First posted 2019-07-09 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Emphysema
Keywords: Lung ultrasound
MeSH Terms: conditions — Pulmonary Emphysema | interventions — Diagnostic Imaging; Respiratory Function Tests; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bullous emphysema: Participants with known bullous emphysema will undergo lung ultrasound according to standard of care clinical practice during a regular follow-up consultation or scheduled hospitalization.
  Interventions: Diagnostic Test: Lung ultrasound; Diagnostic Test: Pulmonary function tests; Other: Clinical examination
- Pneumothorax: Participants hospitalized in pulmonary medicine units for the treatment of a pneumothorax will undergo lung ultrasound according to standard of care clinical practice.
  Interventions: Diagnostic Test: Lung ultrasound; Diagnostic Test: Chest radiography; Other: Clinical examination

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Non-invasive external ultrasonography of the chest wall
Diagnostic Test: Chest radiography — Chest radiography to search for visible pleural edge, synonym with persistent pneumothorax
  Groups: Pneumothorax
Diagnostic Test: Pulmonary function tests — Pulmonary function evaluation as part of routine care for emphysematous patients
  Groups: Bullous emphysema
Other: Clinical examination — Standard clinical examination performed by investigating physician

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a frequent disease affecting a growing number of adults in the world which is responsible for a large public health burden through heavy morbidity and mortality.

Emphysema is one of a wide spectrum of pulmonary complications linked to COPD, defined as the abnormal permanent enlargement of the airspaces distal to the terminal bronchioles accompanied by destruction of the alveolar wall. Disease progression is correlated to worsening and enlargement of emphysema lesions, sometimes conflating in sizeable bullae, deleterious to normal mechanical pulmonary function. Bullous emphysema (BE) is sometimes eligible to invasive curative treatment through surgery or interventional bronchoscopy.

Diagnosis of BE relies on computerized tomodensitometry (CT), the gold-standard for evaluating pulmonary parenchyma. However, CT is not always available, and bullous emphysema can present as pneumothorax on chest radiography.

The practice of lung ultrasound is currently growing in respiratory medicine and emergency departments owing to an increasing amount of evidence showcasing its reliability as a diagnostic tool, most notably for pneumothorax and other pleural diseases. Despite BE having been reported to present similarly to pneumothorax in ultrasound, its characteristics have not yet been precisely described.

The primary aim of this study is to describe BE using lung ultrasound. Participants with known BE on CT will undergo a simple ultrasound examination. The secondary aim is to compare the characteristics of BE to those of pneumothorax using lung ultrasound. To achieve this, a second group of participants with currently treated pneumothorax will also undergo lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Bullous emphysema group

  * Consultation or scheduled hospitalization in a Pulmonary Medicine department
  * Past medical history of emphysema on computerized tomodensitometry dating less than two years
  * Bullous emphysema with subpleural contact of two or more intercostal spaces on tomodensitometry
* Pneumothorax group

  * Hospitalized in a Pulmonary Medicine department for the treatment of a pneumothorax
  * Patent pneumothorax visible on chest x-ray dating less than 24 hours

Exclusion Criteria:

* Bullous emphysema group

  * Current pneumothorax
  * Past medical history of pleurodesis or pleural thickening homolateral to the bullous emphysema
* All patients

  * Organ failure (hemodynamic, neurological, respiratory)
  * Recent thoracic surgery dating less than 7 days with subcutaneous emphysema
  * Minor participant or otherwise deprived of their freedom or their ability to consent freely
  * No affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple Pulmonary Departments in France, in the setting of University Hospitals. All participants fulfilling inclusion criteria will be included.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of various ultrasound signs in the bullous emphysema group, according to a predetermined sonographic evaluation form, following a standardized segmentation of the chest | 2 years
  The following sonographic signs will be investigated :
  * Pleural sliding (presence/absence)
  * Z lines (presence/absence)
  * A line visibility increase (presence/absence)
  * B line (number per field)
  * pulmonary pulse (presence/absence)
  * lung-point (presence/absence)
  * intercostoaeric line thickness (in mm)
  For qualitative signs, the investigators will present proportions Quantitative signs will be reported using means, medians and standard-deviations

SECONDARY OUTCOMES:
Prevalence of various ultrasound signs in the pneumothorax group, according to a predetermined sonographic evaluation form, following a standardized segmentation of the chest | 2 years
  The following sonographic signs will be investigated :
  * Pleural sliding (presence/absence)
  * Z lines (presence/absence)
  * A line visibility increase (presence/absence)
  * B line (number per field)
  * pulmonary pulse (presence/absence)
  * lung-point (presence/absence)
  * intercostoaeric line thickness (in mm)
  For qualitative signs, the investigators will present proportions Quantitative signs will be reported using means, medians and standard-deviations
Statistical comparison of ultrasound characteristics of bullous emphysema and pneumothorax | 2 years
  * Calculation of sensitivity values of lung ultrasound for bullous emphysema for each sonographic sign. Study design prohibits calculation of specificity.
  * A quantitative discrete score will be constructed by enumerating signs which are positive in favor of bullous emphysema, able to discriminate between both diseases. AUC will be calculated. An AUC < 0.75 will be considered as insufficient for establishing lung ultrasound as a diagnostic test for bullous emphysema. An AUC > 0.75 would prompt further studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Medicine, Thoracic Oncology and Respiratory Intensive Care Department, Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Husseini K, Flament T, Laroumagne S, Basille D, Le Brun M, Noel-Savina E, Richard P, Mangiapan G, Artaud-Macari E. Mapping Bullous Emphysema With Lung Ultrasound: A Prospective Multicentre Study. Respirology. 2025 Jul;30(7):633-643. doi: 10.1111/resp.70021. Epub 2025 Mar 9. PMID 40059443